CLINICAL TRIAL: NCT07396350
Title: Autogenous Dentine Derived Barrier Membrane Versus Extended Platelet Rich Fibrin Membrane in Immediate Implant Placement in Posterior Mandible: a 2 Year Follow up
Brief Title: IMMEDIATE IMPLANT With Different Types of Membrane
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R.26.01.96
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Tooth Extraction
Keywords: dental implant

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immediate implant with dentin-derived membrane (Experimental)
  Interventions: Procedure: immediate implant with dentin-derived barrier membrane
- immediate implant with extended platelet rich fibrin membrane (Experimental)
  Interventions: Procedure: immediate implant with eprf membrane

INTERVENTIONS:
Procedure: immediate implant with dentin-derived barrier membrane — immediate implant with dentin-derived barrier membrane with allograft covering any peri-implant defect and jumping gap.
  Arms: immediate implant with dentin-derived membrane
Procedure: immediate implant with eprf membrane — immediate implant with eprf membrane with allograft covering any peri-implant defect and jumping gap.
  Arms: immediate implant with extended platelet rich fibrin membrane

SUMMARY:
Forty patients will be selected from the outpatient's clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Mansoura University for replacement of non-restorable tooth in posterior mandibular area with immediate implants.

ELIGIBILITY:
Eligibility Criteria:

1. Patients aged 18 years and older.
2. Non-restorable mandibular molars requiring extraction and GBR for immediate implant placement.
3. The tooth that required extraction showed no clinical or radiographic signs of acute infection.
4. There was at least 5 mm of available bone between the superior border of the inferior alveolar canal and the root apex.
5. At least 8 mm inter-arch space for the prosthesis.
6. Patients were free of systemic conditions that absolutely contraindicate implant insertion.
7. Patients with good oral hygiene.
8. Patients capable of adhering to the mandated follow-up appointments.

Exclusion Criteria:

1. Tobacco Smokers.
2. Pregnancy.
3. Patients with a history of radiation to the head and neck.
4. Bruxism and parafunctional habits

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Implant stability | 12 months
  The implant stability was evaluated immediately postoperatively and after 3, 6, and 12 months. An Osstell Mentor device (Osstell, Savadaled, Sweden; Integration Diagnostics) was utilized to assess implant stability utilizing resonance frequency analysis (RFA). Measurements were made at 90° in four different directions in order to calculate the RFA value. The implant stability quotient (ISQ) was calculated by averaging the results for each implant.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided